CLINICAL TRIAL: NCT02659891
Title: Immunoglobulin (Privigen®) Therapy to Treat BK Viremia and Prevent Alloimmune Activation in Kidney Transplant Recipients
Brief Title: IVIg to Treat BK Viremia in Kidney Transplant Recipients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Hannah Gilligan, Transplant Nephrologist, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P000224
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplantation; BK Virus; Isoantibodies
MeSH Terms: interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Group 1 (Treatment) (Active Comparator): Intravenous immune globulin (IVIg; Privigen®) 1g/kg monthly for 2 months with immunosuppression reduction.
  Interventions: Biological: IVIg
- Group 2 (Control) (Placebo Comparator): Placebo infusion monthly for 2 months with immunosuppression reduction
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IVIg
  Other Names: Privigen®
  Arms: Group 1 (Treatment)
Other: Placebo
  Arms: Group 2 (Control)

SUMMARY:
The overall goal of this study is to rapidly improve clearance of BK viremia with Immunoglobulin (Privigen®) thereby decreasing the potential for formation of alloantibodies in renal transplant recipients that have had immunosuppression reduction due to BK viremia. Our approach is to perform a prospective, randomized, placebo controlled trial intravenous immune globulin (IVIg; Privigen®) plus protocolized immunosuppression reduction versus placebo and protocolized immunosuppression reduction in patients with BK viremia post-kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Female subject is either postmenopausal for at least 1 year before the screening visit, is surgically sterilized or if they are of childbearing potential, agree to practice effective methods of contraception from the time of signing the informed consent form through 30 days after the last dose of intravenous immune globulin, or agree to completely abstain from heterosexual intercourse.
* Kidney transplant recipients (living and deceased donors) with new onset BK viremia (defined as BKV plasma DNA load >1000 copies/mL by real-time PCR within 2 weeks of enrollment). For values >5000 copies/mL repeat testing is not required. For values ≤5000 copies/mL repeat testing should be performed to confirm viremia before enrollment.
* Immunosuppression therapy at enrollment with tacrolimus, MPA, +/- prednisone.
* Men and Women 18 to 75 years of age.

Exclusion Criteria:

* Absence of a DQ mismatch to the donor.
* Patient had known HLA antibodies directed to the donor antigens (pre-formed DSA) prior to transplant.
* Known to be positive for donor specific anti-HLA antibodies (IgG) at time of enrollment from the most recently drawn sample. (DSA MFI>1000 is considered positive). DSA is detected via center's standard of care testing. If center does not routinely screen then patient may still be enrolled.
* History of biopsy proven acute rejection (cellular or antibody) at any time prior to enrollment.
* BKV plasma DNA viral load >300,000 copies/ml.
* Patient who have received intravenous immune globulin for any reason within 1 month prior to enrollment.
* Patient with an estimated glomerular filtration rate (MDRD) ≤ 30 ml/min at time of study entry.
* Patient with selective IgA deficiency or have known antibodies to IgA.
* Patient with history of hyperprolinemia.
* Patient with a previous history of a severe systemic or anaphylactic response to intravenous immune globulin.
* Female subject is pregnant or lactating.
* Current HCV positivity (by PCR).
* History of HBsAg-positive.
* Patients who are HIV-positive.
* Recipients of a kidney from a donor who tests positive for HIV or HBsAg
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Inability to perform follow-up or to undergo renal allograft biopsy.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-05; Primary Completion 2020-12-10 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
BK Viremia | 3 Months
  Resolution of BK viremia by 3 months post-enrollment. Resolution is defined as a decrease in viral load of BKV in the plasma to <1000 copies/mL.

SECONDARY OUTCOMES:
Donor specific anti-HLA antibodies | 12 Months
  Prevention of new donor specific anti-HLA antibodies (DSA)
Kidney graft survival | 12 Months
Acute Cellular Rejection | 12 Months
  Incidence of acute cellular rejection (Banff 2013 Criteria)
BK Nephropathy | 12 Months
  Proportion of BKV nephropathy
Acute Antibody Mediated Rejection | 12 Months
  Incidence of acute antibody mediated rejection
Interstitial Fibrosis or Transplant Glomerulopathy | 12 Months
  Incidence of interstitial fibrosis or transplant glomerulopathy
Glomerular Filtrition Rate (GFR) | 12 Months
  Proportion of delta decline in estimated glomerular filtration rate (MDRD) of >20%
BKV remission | Up to 24 Months
  Length of BKV remission (time from clearance of BK viremia to reappearance of BK viremia (plasma DNA load >1000 copies/mL x 2 measures that are a 4weeks apart) or end of study

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Gilligan, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts